CLINICAL TRIAL: NCT04611282
Title: Micro and Macrosurgical Treatment of Gingival Recessions: a Randomized Clinical Trial
Brief Title: Surgical Treatment of Gingival Recessions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Medipol University Hospital (Other)
Collaborators: Kocaeli University (Other)
Responsible Party: Principal Investigator, Begum Alkan, Periodontology specialist, Istanbul Medipol University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Mamtograrct
Record Dates: First submitted 2020-10-12; First posted 2020-11-02 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Clinical Trial; Connective Tissue; Gingival Recession; Microsurgery
MeSH Terms: conditions — Gingival Recession

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Microsurgery group (Experimental): All defects were treated with a CPF plus an SCTG by the same investigator using microsurgery technique.
  Interventions: Procedure: surgical techniques in the treatment of localized gingival recession defects.
- Macrosurgery group (Active Comparator): All defects were treated with a CPF plus an SCTG by the same investigator using macrosurgery technique.
  Interventions: Procedure: surgical techniques in the treatment of localized gingival recession defects.

INTERVENTIONS:
Procedure: surgical techniques in the treatment of localized gingival recession defects. — Micro or macrosurgical echniques were performed using a coronally positioned flap with a subepithelial connective tissue graft.

SUMMARY:
The purpose of this study was to compare the effectiveness of microsurgical and macrosurgical approaches on CPFs plus SCTGs for the treatment of localized gingival recession defects (Miller class I or II) over the course of 6 months based on clinical periodontal parameters, periodontal phenotypes, and the postoperative complaints and satisfaction levels of the patients. We hypothesized that root coverage achieved through microsurgery in Miller I or II gingival recessions would improve clinical periodontal outcomes and the periodontal phenotype, with greater postoperative comfort and aesthetic satisfaction in comparison with conventional macrosurgical techniques. Miller Class I and II gingival recession defects, at least 3.0 mm deep, were selected and randomly assigned to receive micro or macrosurgical techniques. Both techniques were performed using a coronally positioned flap with a subepithelial connective tissue graft. Plaque and gingival indices, gingival recession depth and width, probing pocket depth, bleeding on probing, clinical attachment level, width of keratinized gingiva, aesthetic score and percentage of root coverage, postoperative complaints, and satisfaction of the participants completing the study were evaluated at follow-up 1st, 3rd and 6th months.

ELIGIBILITY:
Inclusion Criteria:

-

All participants were:

* adults aged 18 years or over
* systemically and periodontally healthy
* met the eligibility criteria for localized gingival recession of the canine or premolar teeth according to the Miller classification scheme

Exclusion Criteria:

-

Exclusion criteria included the following:

* medical disorders such as diabetes mellitus, immunologic disorders, and hepatitis;
* a history of chemotherapy or radiotherapy;
* a history of alcoholism or drug abuse;
* a history of previous mucogingival surgery at the gingival recession site;
* medications known to affect gingival tissues;
* antibiotic treatment in the past 6 months;
* smoking >10 cigarettes per day for >5 years, and;
* current pregnancy or lactation.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2017-05 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Percentage of root coverage | 6 months
  The primary endpoint for efficacy of the gingival recession was the percentage of root coverage at baseline and 6-months postsurgery, as measured by gingival recession depth.

SECONDARY OUTCOMES:
Changes in Gingival recession depth | 6 months
Changes in Gingival recession width | 6 months
Changes in Keratinized gingival width | 6 months
visual analog scale | 6 months
  A visual analog scale was used to evaluate postoperative complaints regarding the recipient and donor sites according to graft size and postoperative satisfaction values (level of the gingival margin, gingival tissue color, dentin hypersensitivity, and root coverage) during the follow-up period. A 10 cm VAS, with "none" / "unhappy" at the left end and "unbearable" / "happy" at the right end was prepared for each patient.

IPD SHARING:
Plan to Share IPD: No